CLINICAL TRIAL: NCT05905341
Title: A PHASE 1, OPEN-LABEL, MULTICENTER, DOSE ESCALATION AND DOSE EXPANSION STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, PHARMACODYNAMICS, AND ANTITUMOR ACTIVITY OF PF-07224826, AS A SINGLE AGENT AND IN COMBINATION WITH ENDOCRINE THERAPY IN PARTICIPANTS WITH ADVANCED SOLID TUMORS
Brief Title: Study of PF-07224826, as a Single Agent or in Combination With Endocrine Therapy in Participants With Breast Cancer and Other Advanced Solid Tumors.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: This decision was based on business considerations and not due to specific safety reasons or a request from a regulatory authority.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C5331001
Record Dates: First submitted 2023-05-24; First posted 2023-06-15 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer; Ovarian Cancer; Liposarcoma; Non-small Cell Lung Cancer (NSCLC); Endometrial; Solid Tumors
Keywords: cyclin-dependent kinase 2 (CDK2); cyclin-dependent kinase 4 (CDK4); cyclin-dependent kinase 6 (CDK6); hormone receptor positive/human epidermal growth factor receptor 2 negative (HR+/HER2-)
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Liposarcoma; Carcinoma, Non-Small-Cell Lung | interventions — Fulvestrant

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1 Dose Escalation-Dose Level 1 (Experimental): In Part 1, participants with locally recurrent/advanced or metastatic TNBC, platinum resistant ovarian cancer and other advanced solid tumors will receive PF-07224826 as a single agent. Participants with HR-positive HER2-negative advanced or mBC will receive PF-07224826 in combination with endocrine therapy. PF-07224826 will be administered orally, once daily, on a continuous basis.
  Interventions: Drug: PF-07224826; Combination Product: Fulvestrant
- Part 1 Dose Escalation-Dose Level 2 (Experimental): In Part 1, participants with locally recurrent/advanced or metastatic TNBC, platinum resistant ovarian cancer and other advanced solid tumors will receive PF-07224826 as a single agent. Participants with HR-positive HER2-negative advanced or mBC will receive PF-07224826 in combination with endocrine therapy. PF-07224826 will be administered orally, once daily, on a continuous basis.
  Interventions: Drug: PF-07224826; Combination Product: Fulvestrant
- Part 1 Dose Escalation-Dose Level 3 (Experimental): In Part 1, participants with locally recurrent/advanced or metastatic TNBC, platinum resistant ovarian cancer and other advanced solid tumors will receive PF-07224826 as a single agent. Participants with HR-positive HER2-negative advanced or mBC will receive PF-07224826 in combination with endocrine therapy. PF-07224826 will be administered orally, once daily, on a continuous basis.
  Interventions: Drug: PF-07224826; Combination Product: Fulvestrant
- Part 1 Dose Escalation-Dose Level 4 (Experimental): In Part 1, participants with locally recurrent/advanced or metastatic TNBC, platinum resistant ovarian cancer and other advanced solid tumors will receive PF-07224826 as a single agent. Participants with HR-positive HER2-negative advanced or mBC will receive PF-07224826 in combination with endocrine therapy. PF-07224826 will be administered orally, once daily, on a continuous basis.
  Interventions: Drug: PF-07224826; Combination Product: Fulvestrant
- Part 1 Dose Escalation-Dose Level 5 (Experimental): In Part 1, participants with locally recurrent/advanced or metastatic TNBC, platinum resistant ovarian cancer and other advanced solid tumors will receive PF-07224826 as a single agent. Participants with HR-positive HER2-negative advanced or mBC will receive PF-07224826 in combination with endocrine therapy. PF-07224826 will be administered orally, once daily, on a continuous basis.
  Interventions: Drug: PF-07224826; Combination Product: Fulvestrant
- Part 2 - Arm A (Experimental): In Part 2 Arm A, PF-07224826 will be evaluated in combination with fulvestrant in HR positive HER2 negative advanced or mBC participants who have received prior CDK4/6 inhibitor. PF-07224826 will be administered orally, once daily, on a continuous basis.
  Interventions: Drug: PF-07224826; Combination Product: Fulvestrant
- Part 2 - Arm B (Experimental): In Part 2 Arm B, PF-07224826 will be evaluated in combination with fulvestrant in HR-positive HER2-negative locally advanced or mBC participants whose disease has progressed on prior endocrine therapy and is naïve to CDK4/6 inhibitors. PF-07224826 will be administered orally, once daily, on a continuous basis.
  Interventions: Drug: PF-07224826; Combination Product: Fulvestrant

INTERVENTIONS:
Drug: PF-07224826 — Small molecule cell cycle checkpoint inhibitor that targets CDK 2, 4, and 6, to be administered orally.
  Arms: Part 1 Dose Escalation-Dose Level 1
Combination Product: Fulvestrant — Competitive ER antagonist, to be administered by intramuscular injection (prefilled syringe).
  Arms: Part 1 Dose Escalation-Dose Level 1
Drug: PF-07224826 — Small molecule cell cycle checkpoint inhibitor that targets CDK 2, 4, and 6, to be administered orally.
  Arms: Part 1 Dose Escalation-Dose Level 2
Combination Product: Fulvestrant — Competitive ER antagonist, to be administered by intramuscular injection (prefilled syringe).
  Arms: Part 1 Dose Escalation-Dose Level 2
Drug: PF-07224826 — Small molecule cell cycle checkpoint inhibitor that targets CDK 2, 4, and 6, to be administered orally.
  Arms: Part 1 Dose Escalation-Dose Level 3
Combination Product: Fulvestrant — Competitive ER antagonist, to be administered by intramuscular injection (prefilled syringe).
  Arms: Part 1 Dose Escalation-Dose Level 3
Drug: PF-07224826 — Small molecule cell cycle checkpoint inhibitor that targets CDK 2, 4, and 6, to be administered orally.
  Arms: Part 1 Dose Escalation-Dose Level 4
Combination Product: Fulvestrant — Competitive ER antagonist, to be administered by intramuscular injection (prefilled syringe).
  Arms: Part 1 Dose Escalation-Dose Level 4
Drug: PF-07224826 — Small molecule cell cycle checkpoint inhibitor that targets CDK 2, 4, and 6, to be administered orally.
  Arms: Part 1 Dose Escalation-Dose Level 5
Combination Product: Fulvestrant — Competitive ER antagonist, to be administered by intramuscular injection (prefilled syringe).
  Arms: Part 1 Dose Escalation-Dose Level 5
Drug: PF-07224826 — Small molecule cell cycle checkpoint inhibitor that targets CDK 2, 4, and 6, to be administered orally.
  Arms: Part 2 - Arm A
Combination Product: Fulvestrant — Competitive ER antagonist, to be administered by intramuscular injection (prefilled syringe).
  Arms: Part 2 - Arm A
Drug: PF-07224826 — Small molecule cell cycle checkpoint inhibitor that targets CDK 2, 4, and 6, to be administered orally.
  Arms: Part 2 - Arm B
Combination Product: Fulvestrant — Competitive ER antagonist, to be administered by intramuscular injection (prefilled syringe).
  Arms: Part 2 - Arm B

SUMMARY:
This is a Phase 1, open-label, multicenter, dose escalation and dose expansion study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and antitumor activity of PF-07224826, as a single agent or in combination with endocrine therapy in participants with advanced solid tumors. This study will be divided into dose escalation/finding (Part 1) and dose expansion (Part 2).

In Part 1, participants with locally recurrent/advanced or metastatic Triple Negative Breast Cancer (TNBC), platinum resistant ovarian cancer and other advanced solid tumors will receive PF-07224826 as a single agent. Participants with HR-positive HER2-negative advanced or mBC will receive PF-07224826 in combination with endocrine therapy.

In Part 2 (Arm A), PF-07224826 will be evaluated in combination with fulvestrant in HR-positive HER2-negative advanced or mBC participants who have received prior CDK4/6 inhibitor. In Part 2 (Arm B), PF-07224826 will be evaluated in combination with fulvestrant in HR-positive HER2-negative locally advanced or mBC participants whose disease has progressed on prior endocrine therapy and is naïve to CDK4/6 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Part 1:

  * Participants with HR-positive HER2-negative locally advanced or metastatic breast cancer.
  * Participants with locally recurrent/advanced or metastatic TNBC.
  * Participants with advanced platinum resistant epithelial ovarian cancer (EOC)/fallopian tube cancer/primary peritoneal cancer (PPC).
  * Other advanced solid tumor types: Tumors other than BC or Ovarian: NSCLC, prostate, endometrial, liposarcoma, or other tumors with cyclin D (CCND) and cyclin E (CCNE) implicated in pathogenesis either by gene amplification or overexpression.
* Part 2 (Arm A): Participants with HR positive HER2 negative locally advanced or mBC (post CDK4/6 inhibitors).
* Part 2 (Arm B): Participants with HR positive HER2 negative locally advanced or mBC (naïve to CDK4/6 inhibitors).
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1.
* Adequate Bone Marrow Function

Exclusion Criteria:

* Known active uncontrolled or symptomatic central nervous system (CNS) metastases, carcinomatous meningitis, or leptomeningeal disease as indicated by clinical symptoms, Cerebral edema, and/or progressive growth. Participants with a history of CNS metastases or cord compression are eligible if they have been definitively treated (eg, radiotherapy, stereotactic surgery) and are clinically stable off anticonvulsants and steroids for at least 4 weeks before enrollment and have no evidence of progression at time of study enrollment.
* Participants with advanced/metastatic, symptomatic, visceral spread, that are at risk of life-threatening complications in the short term (eg, including participants with massive uncontrolled effusions [pleural, pericardial, peritoneal], pulmonary lymphangitis, and over 50% liver involvement).
* Any other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ.
* Last anticancer treatment within 2 weeks (or 5 half-lives, whichever is shorter), unless the last immediate anticancer treatment contained an antibody-based agent(s) (approved or investigational), then the interval of 4 weeks or 5 half-lives (whichever is shorter) is required prior to receiving the study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2026-04-14 (Estimated); Study Completion 2028-04-13 (Estimated)

PRIMARY OUTCOMES:
Part 1: First cycle dose limiting toxicities (DLTs) | Cycle 1 (28 days)
Part 1 and Part 2: Adverse events (AEs) as characterized by type, frequency, severity (as graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v 5.0), timing, seriousness and relationship to study therapy. | From the first dose to earliest of 28 days post last dosing date or day of new anticancer therapy -1 day.
Part 1 and Part 2: Number of participants with Clinical Laboratory abnormalities | From the first dose to earliest of 28 days post last dosing date or day of new anticancer therapy -1 day.
Part 1 and Part 2: Incidence of clinically significant abnormal vital signs. | From the first dose to earliest of 28 days post last dosing date or day of new anticancer therapy -1 day.
Part 2: Preliminary antitumor activity measure for efficacy includes ORR, as assessed using RECIST version 1.1. | From baseline until the date of first documented progression, or date of death of any cause, or date of withdrawal of consent, or date of lost to follow-up, whichever came first.
Part 1 and Part 2: Incidence of clinically significant abnormal ECGs. | From the first dose to earliest of 28 days post last dosing date or day of new anticancer therapy -1 day.

SECONDARY OUTCOMES:
Part1 and Part 2: Maximum Observed Plasma Concentration (Cmax); Single Dose (SD) | Cycle 1 (Pre-dose, Day 1, 8, and 15) and Cycle 2 (Day 1). Each cycle is 28 days.
Part 1 and Part 2: Time to Reach Maximum Observed Plasma Concentration (Tmax); Single Dose (SD) | Cycle 1 (Pre-dose, Day 1, 8, and 15) and Cycle 2 (Day 1). Each cycle is 28 days.
Part 1: Area under the concentration-time curve from 0 to time of last measurable concentration (AUClast) | Cycle 1 (Pre-dose, Day 1, 8, and 15) and Cycle 2 (Day 1). Each cycle is 28 days.
Part 1 and Part 2: Maximum Observed Plasma concentration (Cmax,ss), steady state | Cycle 1 (Pre-dose, Day 1, 8, and 15) and Cycle 2 (Day 1). Each cycle is 28 days.
Part 1 and Part 2: Time to Reach Maximum Observed Plasma Concentration steady state (Tmax, ss) | Cycle 1 (Pre-dose, Day 1, 8, and 15) and Cycle 2 (Day 1). Each cycle is 28 days.
Part 1 and Part 2: Minimum Observed Plasma Concentration (Cmin, ss), steady state | Cycle 1 (Pre-dose, Day 1, 8, and 15) and Cycle 2 (Day 1). Each cycle is 28 days.
Part 1: Area Under the concentration-time curve from 0 to time the end of the dosing interval (AUCtau,ss), steady state | Cycle 1 (Pre-dose, Day 1, 8, and 15) and Cycle 2 (Day 1). Each cycle is 28 days.
Part 2: Accumulation ratio (Rac) | Cycle 1 (Pre-dose, Day 1, 8, and 15) and Cycle 2 (Day 1). Each cycle is 28 days.
Part 1: Objective Response, as assessed using RECIST version 1.1. | From baseline and up to approximately 24 months
Part 1 and Part 2: Duration of Response (DoR) of PF-07224826 alone or in combination with fulvestrant | From baseline and up to approximately 24 months
Part 1 and Part 2: Progression-Free Survival (PFS) of PF-07224826 alone or in combination with fulvestrant | From baseline and up to approximately 24 months
Part 1 and Part 2: Time to Response (TTR) of PF-07224826 alone or in combination with fulvestrant | From baseline and up to approximately 24 months
Part 2: Overall Survival (OS) of PF-07224826 with fulvestrant | From baseline and up to approximately 24 months
Part 2: Clinical benefit response (CBR) of PF-07224826 with fulvestrant | From baseline and up to approximately 24 months
Part 1 and Part 2: Expression of Pharmacodynamic (PD) biomarkers in tumor tissue | From baseline and up to approximately 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5331001